CLINICAL TRIAL: NCT04067206
Title: The Effects Of White Noise, Recorded Mother's Voice, And Minimuffs (Earmuff) On Pain And Comfort In Premature Infants During Heel Lance: Randomized Clinical Trial
Brief Title: The Effects Of Auditory Interventions On Pain And Comfort In Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ayşe Kahraman, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17HEF001
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Premature Birth; Premature Infant
Keywords: Premature; Pain; Comfort; Auditory Interventions
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Intervention Model Description: This experimental study is a randomized controlled research. The infants were randomly assigned to four groups. Three interventions, each alone and in combination, are evaluated in parallel against a control group
Masking Description: The infants were randomly assigned to four groups: i) white noise , ii) recorded mother's voice, iii) MiniMuffs, and iv) control. Masking could not be performed because the mother's voice was requested from the mothers.Masking could not be done because researchers and observers heard the mother's voice and white noise and saw the mimimuff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Recorded mothers' voice group. (Experimental): The mothers of the babies were given voice recorders and asked to record their voice in a comfortable room saying whatever they wanted to their baby. Each mother recorded her voice for 3-5 minutes. The voice recorder was placed at the baby's foot five minutes before the procedure and then played to the baby during the procedure.The sound level was adjusted to 50 decibels using the Benetech Digital Sound Level Meter for the mother's voice and white noise groups.
  Interventions: Other: RECORDED MOTHER'S VOICE
- White Noise (Experimental): The white noise was started five minutes before the heel lance and was played to the baby during the procedure. Dr. Harvery Karp's "The Happiest Baby," which consists of only intrauterine sounds, was used. The speakers were placed at a distance of about 30 cm from the foot of the neonate. The sound level was adjusted to 50 decibels using the Benetech Digital Sound Level Meter for the mother's voice and white noise groups.
  Interventions: Other: White Noise
- MiniMuffs (Experimental): MiniMuffs placed on their ears five minutes before the procedure to reduce the environmental noise. Latus MiniMuffs - Neonatal Noise Attenuators have been developed for newborns and premature babies. MiniMuffs protect the sensitive ears of the premature and provide a safe environment for healthy development.
  Interventions: Other: MiniMuff
- Control Group (No Intervention): The control group who were administered standard care.

INTERVENTIONS:
Other: RECORDED MOTHER'S VOICE — The mothers of the babies were given voice recorders and asked to record their voice in a comfortable room saying whatever they wanted to their baby. Each mother recorded her voice for 3-5 minutes. The voice recorder was placed at the baby's foot five minutes before the procedure and then played to the baby during the procedure.The sound level was adjusted to 50 decibels using the Benetech Digital Sound Level Meter for the mother's voice and white noise groups.
  Arms: Recorded mothers' voice group.
Other: White Noise — The white noise was started five minutes before the heel lance and was played to the baby during the procedure. Dr. Harvery Karp's "The Happiest Baby," which consists of only intrauterine sounds, was used. The speakers were placed at a distance of about 30 cm from the foot of the neonate. The sound level was adjusted to 50 decibels using the Benetech Digital Sound Level Meter for the mother's voice and white noise groups.
  Arms: White Noise
Other: MiniMuff — MiniMuffs placed on their ears five minutes before the procedure to reduce the environmental noise. Latus MiniMuffs - Neonatal Noise Attenuators have been developed for newborns and premature babies. MiniMuffs protect the sensitive ears of the premature and provide a safe environment for healthy development.
  Arms: MiniMuffs

SUMMARY:
This study investigated the effects of three interventions -recorded mother's voice, white noise, and MiniMuffs, muffs used to attenuate environmental sounds- applied during a heel lance on pain and comfort in premature infants. This randomized controlled research was conducted in a state hospital tertiary-level neonatal intensive care unit. Sixty-four premature neonates with a gestational age of 31-36 who were stable, didn't receive mechanic ventilation and has been started feeding participated. The infants were randomly assigned to four groups: i) white noise , ii) recorded mother's voice, iii) MiniMuffs (earmuff), and iv) control. Five minutes before the procedure the white noise and mother's voice played and MiniMuffs placed on babies' ears. The heel lance procedure was recorded on a camera. The camera recordings were evaluated for premature infants' pain and comfort according to the Neonatal Infant Pain Scale (NIPS) and the Comfort behavior (COMFORTneo) scale.

DETAILED DESCRIPTION:
Auditory interventions are commonly used during procedural analgesic administration in premature neonates. This study investigated the effects of three interventions -recorded mother's voice, white noise, and MiniMuffs, muffs used to attenuate environmental sounds- applied during a heel lance on pain and comfort in premature infants. This experimental study is a randomized controlled research. The data for the research were collected between September 2017 - April 2019. The sample comprised 64 premature infants with gestational ages of 31-36 weeks, who had been hospitalized at the Neonatal Intensive Cate Units (NICU). All infants in the study were in their first postnatal week. The study routine included a heel lance procedure to determine the level of bilirubin and hematocrit. The heel lance was performed with a lancet and the blood was transferred to the hematocrit pipette. All heel lances were conducted by the same nurse. Power analysis was conducted to determine the number of samples needed. Predicting that the NIPS score would decrease by 30-35% and decrease from 6 to 4-4.5 with 0.05 error and 80% power, the intervention groups yielded 64 infants divided into four groups of 16 as the target sample number. 80 infants included in the study, taking into account the loss of sample. Sixteen infants were excluded from the study. Sixty-four premature infants submitted for heel lance were evaluated.The randomization list was prepared by a third person using R version 3.1.3 package program and considering the gender factor. The list was concealed from the researcher and the family of the baby, and it was given to the researcher only during the procedure. The infants were randomly assigned to four groups. The infants were randomly assigned to four groups: i) white noise , ii) recorded mother's voice, iii) MiniMuffs, and iv) control. Five minutes before the procedure the white noise and mother's voice played and MiniMuffs placed on babies' ears. Heel lance procedures were recorded with a camera. Camera recording started before the procedure and continued until the baby stopped crying. The videos evaluated independently by two scientists (observers) who were specialists in neonatal services and pain. Observers evaluated infants' comfort, pain, and distress based on NIPS and COMFORTneo. In order to evaluate the agreement between the observers for the total scores of NIPS and COMFORTneo, pain estimation, and distress estimation, intraclass correlation coefficient were determined.

ELIGIBILITY:
Inclusion Criteria:

* Born by cesarean section
* Non-supported by a mechanical ventilator or NCPAP
* Started to feed
* Within the first 10 days of postnatal

Exclusion Criteria:

* Had a major congenital malformation,
* Apgar score was less than 5 in the 1st-minute and less than 7 in the 5th-minute
* Received a sedative, muscle relaxant, corticosteroid, or analgesic therapy,
* First blood sampling attempt was unsuccessful
* MiniMuffs moved from their ears during the procedure
* Mothers who had problems recording their voice.

Ages: 31 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2019-04-13 (Actual)

PRIMARY OUTCOMES:
Pain (Neonatal Infant Pain Scale-NIPS) | During procedure
  Neonatal Infant Pain Scale: The Neonatal Infant Pain Scale (NIPS), developed by Lawrence et al. (1993), is a behavioral scale and can be used with both full-term and preterm infants. The Cronbach's alpha coefficients of the scale were 0.95, 0.87, and 0.88 before, during, and after the procedure, respectively. In NIPS, five behavioral indicators (facial expression, cry, arms, legs, and state of arousal) and one physiological parameter (breathing pattern) are assessed. Each behavioral indicator is scored with 0 or 1 except "cry", which has three descriptors (scored with a 0, 1, or 2). The total pain score ranges between 0 and 7 with 0-2 points indicating mild to no pain, 3-4 indicating mild to moderate pain, and >4 indicating severe pain.
COMFORT (COMFORTneo Scale) | during procedure
  The COMFORTneo scale is a Likert-type scale consisting of seven parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tonus. As well as determining comfort, the COMFORTneo scale is a tool that includes the Numerical Assessment Scales, which allow nurses to assess the pain and distress of the baby. "Respiratory response" and "crying" scores were recorded from the infants connected to mechanical ventilators and spontaneously breathing infants, respectively. The lowest score on the scale is 6 and the highest is 30. If the total score of the scale is between 14-30, the baby has pain or distress, is uncomfortable, and needs intervention to provide comfort. In addition, 4-6 points from the Numerical Assessment Scales indicates moderate and 7-10 points indicates severe pain and distress.The validity and reliability study of the Turkish version of the scale was conducted. Cronbach's alpha coefficient of the scale was 0.82-0.92.

SECONDARY OUTCOMES:
Heart rates | heart rate values recorded 5 minutes and 1 minute before the procedure, during the procedure, and 1 minute and 5 minutes after the procedure.
  Heart rates were monitored using Pulse Oximetry and were video-recorded.
Crying time | during procedure
  Crying duration was noted by watching video recordings.
the oxygen saturation | oxygen saturation values recorded 5 minutes and 1 minute before the procedure, during the procedure, and 1 minute and 5 minutes after the procedure.
  oxygen saturation was monitored using Pulse Oximetry and were video-recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zümrüt Başbakkal, Professor, Study Director — Ege University
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are unknown and will be made available at a later date.

REFERENCES:
- [Background] Chirico G, Cabano R, Villa G, Bigogno A, Ardesi M, Dioni E. Randomised study showed that recorded maternal voices reduced pain in preterm infants undergoing heel lance procedures in a neonatal intensive care unit. Acta Paediatr. 2017 Oct;106(10):1564-1568. doi: 10.1111/apa.13944. Epub 2017 Jul 5. PMID 28580602
- [Background] Kucukoglu S, Aytekin A, Celebioglu A, Celebi A, Caner I, Maden R. Effect of White Noise in Relieving Vaccination Pain in Premature Infants. Pain Manag Nurs. 2016 Dec;17(6):392-400. doi: 10.1016/j.pmn.2016.08.006. Epub 2016 Oct 15. PMID 27751753